CLINICAL TRIAL: NCT03068299
Title: Effects of Music and Dance on Cognition, Frailty, and Burden in Elderly Caregivers Living in Rural Communities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Allan Gustavo Brigola, Principal Investigator, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 63133316.4.0000.5504
Record Dates: First submitted 2017-02-22; First posted 2017-03-01 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Cognitive Decline; Memory Loss; Frail Elderly Syndrome; Burden, Dependency
Keywords: Prevention; Cognition; Aged care; Caregivers; Frail elderly; Dancing therapy; Rural population
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Intervention Model Description: The dance protocol will be applied to the experimental group (n=29) in the USFs and the control group (n=29) will receive health care, including guidance on health care and practices
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dance (Experimental): n=29 participants randomized. Cognition performance, frailty and burden will be measured at baseline and after of interventions (6 months after baseline). Instruments of measurement described in Time Frame.
  Interventions: Other: Dance
- Health care guidance (Experimental): n=29 participants randomized. Cognition performance, frailty and burden will be measured at baseline and after of interventions (6 months after baseline). Instruments of measurement described in Time Frame.
  Interventions: Other: Health care guidance

INTERVENTIONS:
Other: Dance — Sessions of sixty minutes each, which will take place weekly, totaling 24 weeks (6 months). Ten minutes from the start of each session will be reserved for initial exercises, with movements of the upper limbs, lower, accompanied by a motivational music. The process of identifying and memorizing the movements will be carried out as many times as the group deems necessary. The rhythms include combinations of circular and ballroom dances, including waltz, cha-cha-cha, cancan, among others. In all the sessions, the last fifteen minutes are reserved for a conversation about the dance learned/practiced in the day. It is expected to have reached the proposal of a practice of 15 different choreographies and that this was a pleasant moment for all the participants.
  Arms: Dance
Other: Health care guidance — Control group will receive attention, through guidelines for care and health practices for the caregiver and the elderly care recipient. This attention should occur in the same number of sessions of the dance and group intervention group. The control group should follow the same subdivision of the intervention group, in terms of the number of participants per subgroup. The subjects of the guidelines will be raised by the demand of the participants themselves and then worked in an interdisciplinary way.
  Arms: Health care guidance

SUMMARY:
This research aims to analyze the effects of senior dance on the cognition, frailty, and burden in elderly caregivers of rural communities. This is a randomized clinical trial to be conducted with a sample of 58 elderly caregivers residing in rural communities. Data collection will be performed in the homes of the elderly and/or in the dependencies of the Family Health units (USFs - primary health care systems). They will answer Socio-demographic characterization instrument, ACE-R Battery, and electroencephalography for cognitive evaluation, five Fragility criteria proposed by Fried et al and Zarit Burden Inventory. The dance protocol will be applied to the experimental group (n=29) in the USFs and the control group (n=29) will receive health care, including guidance on health care and practices. The protocols include 24 interventions, 60 minutes each, weekly, during 6 months. Analysis of effects comparisons will be conducted between groups and be comparing baseline with final measurements. Dance intervention is expected to exert important positive effects on all study variables (cognitive performance, fragility assessment, and caregiver burden), compared to the group. The intervention of the control group is expected to exert positive effects on some variables of the study (mainly, caregiver burden).

DETAILED DESCRIPTION:
Sample Variables above described of 58 participants will be measured. The participants will be randomized to the dance group (experimental) and to the health care guidance group (control). The group will be paired by age, sex, and schooling. This study focused on prevention of cognitive performance decline, frailty and burden.

ELIGIBILITY:
Inclusion Criteria:

1. - Caregivers of elderly registered in Units of Family Health system in rural communities of São Carlos, Brazil.
2. - Over 60 years old.
3. - Living rural area.

Exclusion Criteria:

1 - Sufficient sensory or language difficulties that impede the participation of the intervention and the measurement of the variables

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Effects of dance on cognition performance | Change from Baseline in Addenbrooke's Cognitive Examination at 6 months.
  It is expected Dance exerts important positive effects on cognition performance compared to baseline.
Effects of dance on frailty | Change from Baseline in Fried Frailty Criteria at 6 months.
  It is expected Dance exerts important positive effects on frailty compared to baseline.
Effect of dance on burden | Change from Baseline in Zarit Burden Interview at 6 months.
  It is expected Dance exerts important positive effects on burden compared to baseline.

SECONDARY OUTCOMES:
Effects of HCG on burden | Change from Baseline in Zarit Burden Interview at 6 months.
  It is expected Health Care Guidance (HCG) exerts important positive effects on burden compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Allan G Brigola, Ph.D., Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Federal University of São Carlos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
No participant data will be shared with other research. However, the analyzed results will be published in papers.

REFERENCES:
- Available data/document: Ethics Acceptance letter: 63133316.4.0000.5504 — http://plataformabrasil.saude.gov.br/login.jsf — Enter with number CAAE box (63133316.4.0000.5504) and access the official document of ethics acceptance letter of study.